CLINICAL TRIAL: NCT02528513
Title: Midazolam Used Alone or Sequential Use of Midazolam and Propofol/Dexmedetomidine for Long-Term Sedation in Critically Ill, Mechanically Ventilated Patients: a Prospective, Randomized Study
Brief Title: Midazolam Used Alone or Sequential Use of Midazolam and Propofol/Dexmedetomidine in Mechanically Ventilated Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yongfang, Zhou Yongfang, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HaxiICU
Record Dates: First submitted 2015-08-15; First posted 2015-08-19 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Mechanical Ventilation; Complication; Delirium
Keywords: sedation; Midazolam; Propofol; Dexmedetomidine
MeSH Terms: conditions — Delirium | interventions — Midazolam; Fentanyl; Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- midazolam (Experimental): 1. Midazolam is started with an infusion bolus of 0.03-0.30 mg/kg and continuous infusion of 0.03-0.20 mg/kg/h, with the dosage adjusted to achieve the desired level of sedation.
  2. After the spontaneous breathing trial safety screen is passed, midazolam will continue to be used for sedation, with the dosage adjusted to achieve the desired level of sedation.
  Interventions: Drug: midazolam; Drug: Fentanyl; Procedure: Procedure:sedation assessment; Procedure: Procedure:Weaning; Drug: midazolam(used for passing the SBT safety screen)
- midazolam/propofol (Experimental): 1. Midazolam is started with an infusion bolus of 0.03-0.30 mg/kg and continuous infusion of 0.03-0.20 mg/kg/h, with the dosage adjusted to achieve the desired level of sedation.
  2. After the spontaneous breathing trial safety screen is passed, midazolam is switched to propofol, which is administered at the maintenance dosage of 0.50-3.00mg/kg/h, with the dosage adjusted to achieve the desired level of sedation.
  Interventions: Drug: midazolam; Drug: Fentanyl; Drug: propofol; Procedure: Procedure:sedation assessment; Procedure: Procedure:Weaning
- midazolam/dexmedetomidine (Experimental): 1. Midazolam is started with an infusion bolus of 0.03-0.30 mg/kg and continuous infusion of 0.03-0.20 mg/kg/h, with the dosage adjusted to achieve the desired level of sedation.
  2. After the spontaneous breathing trial safety screen is passed, midazolam is switched to dexmedetomidine, which is administered at an infusion bolus of 0.5 μg/kg over 10 min (given or not according to patients' condition) and the maintenance dosage of 0.2-0.7ug/kg/h, with the dosage adjusted to achieve the desired level of sedation.
  Interventions: Drug: midazolam; Drug: Fentanyl; Drug: Dexmedetomidine; Procedure: Procedure:sedation assessment; Procedure: Procedure:Weaning

INTERVENTIONS:
Drug: midazolam — Midazolam is started with an infusion bolus of 0.03-0.30 mg/kg and continuous infusion of 0.03-0.20 mg/kg/h, with the dosage adjusted to RASS score (-3 to 0).
  Other Names: Liyuxi
Drug: Fentanyl — Fentanyl is used with bolus dosage of 1-2ug/kg and maintenance dosage of 1-2ug/kg/h, with the dosage adjusted to critical care pain observation tool（CPOT）score(0-1).
Drug: propofol — After the spontaneous breathing trial safety screen is passed, midazolam is switched to propofol, which is administered at the maintenance dosage of 0.50-3.00mg/kg/h, with the dosage adjusted to RASS score (-2 to 0).
  Arms: midazolam/propofol
Drug: Dexmedetomidine — After the spontaneous breathing trial safety screen is passed, midazolam is switched to dexmedetomidine, which is administered at an infusion bolus of 0.5μg/kg over 10 min (given or not according to patients' condition) and the maintenance dosage of 0.2-0.7ug/kg/h, with the dosage adjusted to RASS score (-2 to 0).
  Arms: midazolam/dexmedetomidine
Procedure: Procedure:sedation assessment — The nursing staff continuously monitored the sedation depth and adjusted the dosages of sedative and analgesic drugs to maintain the sedation target level. The sedation depth were assessed and recorded every 4 h (or more frequently when indicated).
Procedure: Procedure:Weaning — the respiratory therapists managed patients with a daily interruption of continuous sedation and the spontaneous breathing trial (SBT) protocols daily.
Drug: midazolam(used for passing the SBT safety screen) — After the spontaneous breathing trial safety screen is passed,in the midazolam group, midazolam will continue to be used for sedation, with the dosage adjusted to RASS score (-2 to 0).
  Other Names: Liyuxi
  Arms: midazolam

SUMMARY:
The purpose of this study was to evaluate effects, safety and cost of midazolam used alone or sequential use of midazolam and propofol/dexmedetomidine for long-term sedation in critically ill, mechanically ventilated patients.

DETAILED DESCRIPTION:
It is well known that sedation is frequently required as a component of compassionate care in critically ill patients. Until now, there is no ideal sedation drug and every sedation drug has its advantage and disadvantage for long-term sedation in critically ill, mechanically ventilated patients. The sequential use of midazolam and propofol for long-term sedation was associated with a faster recovery, earlier extubation, shorter mechanical ventilation time and less cost of total ICU treatment compared with midazolam alone, The protocol was associated with less cost of pharmaceutical sedation compared with propofol alone. But, propofol and midazolam may cause respiratory depression and delirium. Both drugs should be stopped after the patient passed the screen of weaning from mechanical ventilation, then it would induce the stress response and agitation, it would cause prolonged sedation and delay extubation.

Dexmedetomidine is a centrally acting a2-receptor agonist, has less effect on arousability and respiratory depression. The purpose of this study was to evaluate effects, safety and cost of midazolam used alone or sequential use of midazolam and propofol/dexmedetomidine for long-term sedation in critically ill, mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Intubated patients;
2. Age≥18 years old;
3. Anticipated Ventilation and sedation duration of at least 72 hours.

Exclusion Criteria:

1. Allergy to the study drug;
2. suspected pregnancy;
3. gross obesity;
4. Extremely unstable of circulatory system, such as systolic blood pressure less than 90 mm Hg despite plasma volume expansion and continuous infusions of vasopressors before the start of study drug infusion;
5. Uncontrolled abnormal hypertension, such as systolic blood pressure more than 180 mmHg or diastolic more than105 mmHg;
6. Heart rate less than 50 bpm;
7. Second or third degree heart block;
8. moribund state;
9. history of alcoholism or intake of anti-anxiety drugs or hypnotics;
10. chronic renal failure;
11. coma by cranial trauma or neurosurgery or unknown etiology or epileptic state;
12. History of neuromuscular disease;
13. unwillingness to provide informed consent by patients or their authorized surrogates following ICU admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Weaning time | From sedation sequential criteria to extubation, up to 28 days

SECONDARY OUTCOMES:
The pharmaceutical costs of sedation | From sedation drug is used to cessation of sedation up to 28 days.
The total ICU costs | From admitted to ICU until ventilation and participants discharged from ICU, up to 28 days.
The incidence of delirium (patients with diagnosis of delirium/ total patients in each group × 100% ) | From sedation drug is used to cessation of sedation, up to 28 days.
  After the daily interruption of continuous sedation,delirium is assessed by the the confusion assessment method for the diagnosis of delirium in ICU(CAM-ICU). If the patient has the clinical features of 1 and 2, or 3,or 4 in the CAM-ICU, delirium can be diagnosed.
Sedation satisfaction degree (The total time within target sedation level/total evaluation times ×100% ) | From sedation drug is used to cessation of sedation up to 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Y Kang, Dr, Study Chair — Critical Medicine Department,West China Hospital of Sichuan University
Locations (1):
- Department of Critical care medicine of West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhou Y, Yang J, Wang B, Wang P, Wang Z, Yang Y, Liang G, Jing X, Jin X, Zhang Z, Deng Y, Hu C, Liao X, Yin W, Tang Z, Tian Y, Tao L, Kang Y. Sequential use of midazolam and dexmedetomidine for long-term sedation may reduce weaning time in selected critically ill, mechanically ventilated patients: a randomized controlled study. Crit Care. 2022 May 3;26(1):122. doi: 10.1186/s13054-022-03967-5. PMID 35505432